CLINICAL TRIAL: NCT04533737
Title: Efficacy and Safety Comparison of Brodalumab Versus Guselkumab in Adult Subjects With Moderate-to-severe Plaque Psoriasis and Inadequate Response to Ustekinumab
Brief Title: Efficacy and Safety of Brodalumab Compared With Guselkumab in the Treatment of Plaque Psoriasis After Inadequate Response to Ustekinumab
Acronym: COBRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment was terminated early due to delays and slow recruitment that significantly jeopardized the trial timelines. There were no safety concerns related to the early termination of the trial.
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0160-1510; 2019-004099-20 (EudraCT Number); U1111-1283-7584 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-02

CONDITIONS: Plaque Psoriasis; Psoriasis Vulgaris; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab; guselkumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Brodalumab (1.5 mL) and guselkumab (1.0 mL) are in pre-filled syringes and packaged open-label. Dummy injections are used for blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (brodalumab + dummy 1) (Experimental): Participants receive:
  * Brodalumab 210 mg (1.5 ml) at Weeks 0, 1, 2, and then every 2 weeks.
  * Dummy 1 (placebo 1.0 ml) at Weeks 0, 4, and then every 8 weeks.
  Interventions: Biological: Brodalumab; Other: Placebo
- Arm 2 (guselkumab + dummy 2) (Active Comparator): Participants receive:
  * Guselkumab 100 mg (1.0 ml) at Weeks 0, 4, and then every 8 weeks.
  * Dummy 2 (placebo 1.5 ml) at Weeks 0, 1, 2, and then every 2 weeks.
  Interventions: Other: Placebo; Biological: Guselkumab

INTERVENTIONS:
Biological: Brodalumab — Pre-filled syringe with 210 mg brodalumab in 1.5 ml solution for subcutaneous injection
  Other Names: Kyntheum®
  Arms: Arm 1 (brodalumab + dummy 1)
Other: Placebo — The placebo solution is similar to the active guselkumab (Dummy 1) or brodalumab (Dummy 2) solution except that it does not contain any active substance
  Other Names: Dummy 1/Dummy 2
Biological: Guselkumab — Pre-filled syringe with 100 mg guselkumab in 1 ml solution for subcutaneous injection
  Other Names: Tremfya®
  Arms: Arm 2 (guselkumab + dummy 2)

SUMMARY:
The trial investigates the efficacy and safety of brodalumab against guselkumab in treatment for patients with moderate-to-severe plaque psoriasis who still have some remaining symptoms after ustekinumab treatment.

DETAILED DESCRIPTION:
Brodalumab is an anti-interleukin 17 receptor A antibody (IL-17RA) and blocks the inflammatory effects of different IL-17 cytokines (IL-17A, IL-17C, IL-17F, IL-17A/F heterodimer, and IL-17E) in the skin. With increasing availability of novel biologics with new targets, the complexity of choosing the appropriate biologic treatment is ever more challenging for physicians. Therefore, the primary objective of this trial is to compare the efficacy of brodalumab versus guselkumab in adult participants with moderate to severe plaque psoriasis and inadequate response to ustekinumab, thereby providing new scientific information that could support decision making in the clinical setting. The study will run approximately 32 weeks for each participant (including a 2- to 4-weeks screening period and a 28-week treatment period), with the primary endpoint measurement at Week 16. Participants receive subcutaneous injections of brodalumab or guselkumab. Dummy injections are also given, so participants and assessors are unaware of which treatment is given.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a diagnosis of plaque psoriasis for at least 6 months before the first administration of investigational medicinal product (IMP) as determined by the investigator.
* Participant has inadequately controlled plaque psoriasis currently treated with ustekinumab, and fulfils ALL of the following criteria:

  1. Ustekinumab administered at least 3 times at or higher than the approved dose or frequency before randomisation.
  2. IGA ≥2 at screening and baseline.
  3. Absolute PASI >3 at screening and baseline.
* Participant has no evidence of active tuberculosis according to local standard of care for patients requiring initiation of a biologic treatment. Participants with adequately treated latent tuberculosis, according to local guidelines, are eligible.

Key Exclusion Criteria:

* Participant was diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions (e.g. eczema) that would interfere with evaluations of the effect of IMP on plaque psoriasis.
* Participant has clinically important active infections or infestations, chronic, recurrent, or latent infections or infestations, or is immunocompromised (e.g. human immunodeficiency virus).
* Participant has any systemic disease (e.g. renal failure, heart failure, hypertension, liver disease, diabetes, anaemia) considered by the investigator to be clinically significant and uncontrolled.
* Participant has a known history of Crohn's disease.
* Participant has any active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma.
* Participant has a history of malignancy within 5 years, except for treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma.
* Participant has a known history of active tuberculosis.
* Participant has a history of suicidal behaviour (i.e. 'actual suicide attempt', 'interrupted attempt', 'aborted attempt', or 'preparatory acts or behaviour') based on the Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire at screening or baseline.
* Participant has any suicidal ideation of severity 4 or 5 ('some intent to act, no plan' or 'specific plan and intent') based on the C-SSRS questionnaire at screening or baseline.
* Participant has a Patient Health Questionnaire-8 (PHQ-8) score of ≥10, corresponding to moderate to severe depression at screening or baseline.
* Participant has previously been treated with any anti-interleukin (IL)-17A, anti-IL 17 receptor subunit A, or anti-IL-23 besides ustekinumab.
* Participant has known or suspected hypersensitivity to any component(s) of the IMPs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (61):
- Austria (2):
  - LEO Pharma Investigational Site, Graz, Styria
  - LEO Pharma Investigational Site, Vienna
- Belgium (3):
  - LEO Pharma Investigational Site, Brussels
  - LEO Pharma Investigational Site, Herstal
  - LEO Pharma Investigational Site, Namur
- Denmark (3):
  - LEO Pharma Investigational Site, Copenhagen
  - LEO Pharma Investigational Site, Hellerup
  - LEO Pharma Investigational Site, Roskilde
- France (8):
  - LEO Pharma Investigational Site, Marseille, Bouches-du-Rhône
  - LEO Pharma Investigational Site, Martigues, Bouches-du-Rhône
  - LEO Pharma Investigational Site, Rouen, Seine-Maritime 10
  - LEO Pharma Investigational Site, Saint-Mandé, Val-de-Marne
  - LEO Pharma Investigational Site, Antony
  - LEO Pharma Investigational Site, Nice
  - LEO Pharma Investigational Site, Saint-Priest-en-Jarez
  - LEO Pharma Investigational Site, Toulouse
- Germany (18):
  - LEO Pharma Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - LEO Pharma Investigational Site, Aachen
  - LEO Pharma Investigational Site, Augsburg
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Bonn
  - LEO Pharma Investigational Site, Bramsche
  - LEO Pharma Investigational Site, Buxtehude
  - LEO Pharma Investigational Site, Cologne
  - LEO Pharma Investigational Site, Darmstadt
  - LEO Pharma Investigational Site, Erlangen
  - LEO Pharma Investigational Site, Frankfurt am Main
  - LEO Pharma Investigational Site, Hamburg
  - LEO Pharma Investigational Site, Kiel
  - LEO Pharma Investigational Site, Mainz
  - LEO Pharma Investigational Site, Memmingen
  - LEO Pharma Investigational Site, Munich
  - LEO Pharma Investigational Site, Münster
  - LEO Pharma Investigational Site, Selters
- Greece (5):
  - LEO Pharma Investigational Site 1, Athens
  - LEO Pharma Investigational Site 2, Athens
  - LEO Pharma Investigational Site 1, Thessaloniki
  - LEO Pharma Investigational Site 2, Thessaloniki
  - LEO Pharma Investigational Site, Thessaloniki
- Italy (4):
  - LEO Pharma Investigational Site, Napoli
  - LEO Pharma Investigational Site, Pisa
  - LEO Pharma Investigational Site, Roma
  - LEO Pharma Investigational Site, Rozzano
- Netherlands (3):
  - LEO Pharma Investigational Site, Bergen op Zoom, Bergen
  - LEO Pharma Investigational Site, Almere Stad, RL Almere
  - LEO Pharma Investigational Site, Amsterdam
- Spain (8):
  - LEO Pharma Investigational Site, Mieres, Principality of Asturias
  - LEO Pharma Investigational Site, Bilbao, Vizcaya
  - LEO Pharma Investigational Site, Alicante
  - LEO Pharma Investigational Site, Barcelona
  - LEO Pharma Investigational Site, Granada
  - LEO Pharma Investigational Site, Madrid
  - LEO Pharma Investigational Site, Pontevedra
  - LEO Pharma Investigational Site, Valencia
- LEO Pharma Investigational Site, Solna, Stockholm County, Sweden
- Switzerland (2):
  - LEO Pharma Investigational Site, Sankt Gallen
  - LEO Pharma Investigational Site, Zurich
- United Kingdom (4):
  - LEO Pharma Investigational Site, Bath, Avon
  - LEO Pharma Investigational Site, Dudley, West Midlands
  - LEO Pharma investigational site, Leeds, West Yorkshire
  - LEO Pharma Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reich K, Bianchi L, Khemis A, Maul JT, Tsianakas A, Schempp CM, Petersen K, Noergaard MM, Puig L. Brodalumab Versus Guselkumab in Patients with Moderate-to-Severe Psoriasis with an Inadequate Response to Ustekinumab: A Randomized, Multicenter, Double-Blind Phase 4 Trial (COBRA). Dermatol Ther (Heidelb). 2024 Feb;14(2):453-468. doi: 10.1007/s13555-023-01092-x. Epub 2024 Feb 1. PMID 38300408

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Brodalumab + Dummy 1): Participants receive:
  * Brodalumab 210 mg (1.5 ml) at Weeks 0, 1, 2, and then every 2 weeks.
  * Dummy 1 (placebo 1.0 ml) at Weeks 0, 4, and then every 8 weeks.
  Brodalumab: Pre-filled syringe with 210 mg brodalumab in 1.5 ml solution for subcutaneous injection.
  Placebo: The placebo solution is similar to the active guselkumab solution except that it does not contain any active substance.
- Arm 2 (Guselkumab + Dummy 2): Participants receive:
  * Guselkumab 100 mg (1.0 ml) at Weeks 0, 4, and then every 8 weeks.
  * Dummy 2 (placebo 1.5 ml) at Weeks 0, 1, 2, and then every 2 weeks.
  Guselkumab: Pre-filled syringe with 100 mg guselkumab in 1 ml solution for subcutaneous injection.
  Placebo: The placebo solution is similar to the active brodalumab solution except that it does not contain any active substance.
Period: Overall Study
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Started | 56 | 57
Completed | 50 | 50
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Population: ITT: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2) | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 48 | 101
  >=65 years | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (10.7) | 51.1 (13.6) | 49.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 40 | 41 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 53 | 53 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 57 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 3 | 5
  Switzerland | 3 | 1 | 4
  Spain | 6 | 10 | 16
  Greece | 6 | 2 | 8
  Netherlands | 1 | 0 | 1
  Sweden | 1 | 2 | 3
  Belgium | 0 | 4 | 4
  Denmark | 0 | 1 | 1
  Italy | 3 | 2 | 5
  France | 11 | 15 | 26
  Germany | 23 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: Having Psoriasis Area and Severity Index (PASI) 100 Response at Week 16
Description: Having 100% improvement from baseline in PASI score. The outcome measure is summarized using the least squares mean percentage of subjects having PASI 100 response at Week 16, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline PASI score.
  The PASI is the most widely used tool in clinical practice and clinical trials to assess psoriasis severity and extent. Assessment is done based on the condition of the disease at the time of evaluation, not in relation to the condition at a previous visit. The investigator assesses the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions (head/neck, trunk, upper extremities, lower extremities) according to a severity scale. The investigator also assesses the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe/extensive condition.
Time Frame: Week 16
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of subjects | 53.4 [40.0 to 66.8] | 35.9 [23.0 to 48.7]

2. Secondary Outcome: Time to PASI 100 Response (Summarized as the Cumulative Incidence for Achieving PASI 100 at Each Timepoint, Stratified by Weight)
Description: Time to having 100% improvement from baseline in PASI score. The outcome measure summarizes the cumulative percentage of subjects with PASI 100 response (stratified by weight) over time, based on the Aalen-Johansen estimator.
  The PASI is the most widely used tool in clinical practice and clinical trials to assess psoriasis severity and extent. Assessment is done based on the condition of the disease at the time of evaluation, not in relation to the condition at a previous visit. The investigator assesses the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions (head/neck, trunk, upper extremities, lower extremities) according to a severity scale. The investigator also assesses the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe/extensive condition.
Time Frame: up to 28 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of subjects
  <=100 kg Week 1: number analyzed (Participants) | 44 | 43
  <=100 kg Week 1 | 0 [0 to 0] | 0 [0 to 0]
  <=100 kg Week 2: number analyzed (Participants) | 44 | 43
  <=100 kg Week 2 | 4.5 [0.8 to 13.7] | 0 [0 to 0]
  <=100 kg Week 4: number analyzed (Participants) | 44 | 43
  <=100 kg Week 4 | 22.7 [11.7 to 36.0] | 2.3 [0.2 to 10.7]
  <=100 kg Week 6: number analyzed (Participants) | 44 | 43
  <=100 kg Week 6 | 34.1 [20.5 to 48.1] | 14.0 [5.6 to 26.1]
  <=100 kg Week 8: number analyzed (Participants) | 44 | 43
  <=100 kg Week 8 | 40.9 [26.3 to 55.0] | 23.3 [11.9 to 36.8]
  <=100 kg Week 10: number analyzed (Participants) | 44 | 43
  <=100 kg Week 10 | 45.5 [30.2 to 59.5] | 27.9 [15.4 to 41.8]
  <=100 kg Week 12: number analyzed (Participants) | 44 | 43
  <=100 kg Week 12 | 61.4 [45.1 to 74.1] | 27.9 [15.4 to 41.8]
  <=100 kg Week 14: number analyzed (Participants) | 44 | 43
  <=100 kg Week 14 | 61.4 [45.1 to 74.1] | 30.2 [17.2 to 44.3]
  <=100 kg Week 16: number analyzed (Participants) | 44 | 43
  <=100 kg Week 16 | 63.6 [47.4 to 76.1] | 39.5 [24.9 to 53.8]
  <=100 kg Week 18: number analyzed (Participants) | 44 | 43
  <=100 kg Week 18 | 63.6 [47.4 to 76.1] | 46.5 [31.0 to 60.6]
  <=100 kg Week 20: number analyzed (Participants) | 44 | 43
  <=100 kg Week 20 | 65.9 [49.6 to 78.0] | 46.5 [31.0 to 60.6]
  <=100 kg Week 22: number analyzed (Participants) | 44 | 43
  <=100 kg Week 22 | 65.9 [49.6 to 78.0] | 46.5 [31.0 to 60.6]
  <=100 kg Week 24: number analyzed (Participants) | 44 | 43
  <=100 kg Week 24 | 68.2 [51.9 to 80.0] | 46.5 [31.0 to 60.6]
  <=100 kg Week 26: number analyzed (Participants) | 44 | 43
  <=100 kg Week 26 | 68.2 [51.9 to 80.0] | 46.5 [31.0 to 60.6]
  <=100 kg Week 28: number analyzed (Participants) | 44 | 43
  <=100 kg Week 28 | 70.5 [54.2 to 81.9] | 48.8 [33.1 to 62.8]
  >100 kg Week 1: number analyzed (Participants) | 12 | 13
  >100 kg Week 1 | 0 [0 to 0] | 0 [0 to 0]
  >100 kg Week 2: number analyzed (Participants) | 12 | 13
  >100 kg Week 2 | 8.3 [0.4 to 32.3] | 0 [0 to 0]
  >100 kg Week 4: number analyzed (Participants) | 12 | 13
  >100 kg Week 4 | 25.0 [5.5 to 51.6] | 0 [0 to 0]
  >100 kg Week 6: number analyzed (Participants) | 12 | 13
  >100 kg Week 6 | 25.0 [5.5 to 51.6] | 7.7 [0.4 to 30.3]
  >100 kg Week 8: number analyzed (Participants) | 12 | 13
  >100 kg Week 8 | 41.7 [14.1 to 67.6] | 7.7 [0.4 to 30.3]
  >100 kg Week 10: number analyzed (Participants) | 12 | 13
  >100 kg Week 10 | 50.0 [19.2 to 74.7] | 15.4 [2.2 to 39.8]
  >100 kg Week 12: number analyzed (Participants) | 12 | 13
  >100 kg Week 12 | 50.0 [19.2 to 74.7] | 15.4 [2.2 to 39.8]
  >100 kg Week 14: number analyzed (Participants) | 12 | 13
  >100 kg Week 14 | 58.3 [24.8 to 81.2] | 23.1 [5.1 to 48.5]
  >100 kg Week 16: number analyzed (Participants) | 12 | 13
  >100 kg Week 16 | 58.3 [24.8 to 81.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 18: number analyzed (Participants) | 12 | 13
  >100 kg Week 18 | 58.3 [24.8 to 81.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 20: number analyzed (Participants) | 12 | 13
  >100 kg Week 20 | 58.3 [24.8 to 81.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 22: number analyzed (Participants) | 12 | 13
  >100 kg Week 22 | 58.3 [24.8 to 81.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 24: number analyzed (Participants) | 12 | 13
  >100 kg Week 24 | 66.7 [30.2 to 87.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 26: number analyzed (Participants) | 12 | 13
  >100 kg Week 26 | 66.7 [30.2 to 87.2] | 30.8 [8.8 to 56.5]
  >100 kg Week 28: number analyzed (Participants) | 12 | 13
  >100 kg Week 28 | 66.7 [30.2 to 87.2] | 30.8 [8.8 to 56.5]

3. Secondary Outcome: Time to PASI 90 Response (Summarized as the Cumulative Incidence for Achieving PASI 90 at Each Timepoint, Stratified by Weight)
Description: Time to having 90% improvement from baseline in PASI score. The outcome measure summarizes the cumulative percentage of subjects with PASI 90 response (stratified by weight) over time, based on the Aalen-Johansen estimator.
  The PASI is the most widely used tool in clinical practice and clinical trials to assess psoriasis severity and extent. Assessment is done based on the condition of the disease at the time of evaluation, not in relation to the condition at a previous visit. The investigator assesses the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions (head/neck, trunk, upper extremities, lower extremities) according to a severity scale. The investigator also assesses the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe/extensive condition.
Time Frame: up to 28 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of subjects
  <=100 kg Week 1: number analyzed (Participants) | 44 | 43
  <=100 kg Week 1 | 0 [0 to 0] | 0 [0 to 0]
  <=100 kg Week 2: number analyzed (Participants) | 44 | 43
  <=100 kg Week 2 | 6.8 [1.7 to 16.9] | 0 [0 to 0]
  <=100 kg Week 4: number analyzed (Participants) | 44 | 43
  <=100 kg Week 4 | 27.3 [15.1 to 41.0] | 9.3 [2.9 to 20.3]
  <=100 kg Week 6: number analyzed (Participants) | 44 | 43
  <=100 kg Week 6 | 56.8 [40.8 to 70.0] | 23.3 [11.9 to 36.8]
  <=100 kg Week 8: number analyzed (Participants) | 44 | 43
  <=100 kg Week 8 | 65.9 [49.6 to 78.0] | 34.9 [21.0 to 49.1]
  <=100 kg Week 10: number analyzed (Participants) | 44 | 43
  <=100 kg Week 10 | 68.2 [51.9 to 79.9] | 39.5 [24.9 to 53.8]
  <=100 kg Week 12: number analyzed (Participants) | 44 | 43
  <=100 kg Week 12 | 72.7 [56.6 to 83.7] | 41.9 [26.9 to 56.1]
  <=100 kg Week 14: number analyzed (Participants) | 44 | 43
  <=100 kg Week 14 | 72.7 [56.6 to 83.7] | 44.2 [29.0 to 58.4]
  <=100 kg Week 16: number analyzed (Participants) | 44 | 43
  <=100 kg Week 16 | 75.0 [59.0 to 85.5] | 48.8 [33.1 to 62.8]
  <=100 kg Week 18: number analyzed (Participants) | 44 | 43
  <=100 kg Week 18 | 75.0 [59.0 to 85.5] | 51.2 [35.3 to 65.0]
  <=100 kg Week 20: number analyzed (Participants) | 44 | 43
  <=100 kg Week 20 | 81.8 [66.2 to 90.7] | 55.8 [39.6 to 69.3]
  <=100 kg Week 22: number analyzed (Participants) | 44 | 43
  <=100 kg Week 22 | 81.8 [66.2 to 90.7] | 55.8 [39.6 to 69.3]
  <=100 kg Week 24: number analyzed (Participants) | 44 | 43
  <=100 kg Week 24 | 81.8 [66.2 to 90.7] | 55.8 [39.6 to 69.3]
  <=100 kg Week 26: number analyzed (Participants) | 44 | 43
  <=100 kg Week 26 | 81.8 [66.2 to 90.7] | 55.8 [39.6 to 69.3]
  <=100 kg Week 28: number analyzed (Participants) | 44 | 43
  <=100 kg Week 28 | 81.8 [66.2 to 90.7] | 55.8 [39.6 to 69.3]
  >100 kg Week 1: number analyzed (Participants) | 12 | 13
  >100 kg Week 1 | 0 [0 to 0] | 0 [0 to 0]
  >100 kg Week 2: number analyzed (Participants) | 12 | 13
  >100 kg Week 2 | 16.7 [2.4 to 42.4] | 7.7 [0.4 to 30.3]
  >100 kg Week 4: number analyzed (Participants) | 12 | 13
  >100 kg Week 4 | 33.3 [9.4 to 60.0] | 15.4 [2.2 to 39.8]
  >100 kg Week 6: number analyzed (Participants) | 12 | 13
  >100 kg Week 6 | 58.3 [25.1 to 81.1] | 23.1 [5.1 to 48.5]
  >100 kg Week 8: number analyzed (Participants) | 12 | 13
  >100 kg Week 8 | 58.3 [25.1 to 81.1] | 23.1 [5.1 to 48.5]
  >100 kg Week 10: number analyzed (Participants) | 12 | 13
  >100 kg Week 10 | 58.3 [25.1 to 81.1] | 23.1 [5.1 to 48.5]
  >100 kg Week 12: number analyzed (Participants) | 12 | 13
  >100 kg Week 12 | 58.3 [25.1 to 81.1] | 23.1 [5.1 to 48.5]
  >100 kg Week 14: number analyzed (Participants) | 12 | 13
  >100 kg Week 14 | 66.7 [30.8 to 87.0] | 30.8 [8.8 to 56.5]
  >100 kg Week 16: number analyzed (Participants) | 12 | 13
  >100 kg Week 16 | 66.7 [30.8 to 87.0] | 46.2 [17.9 to 70.7]
  >100 kg Week 18: number analyzed (Participants) | 12 | 13
  >100 kg Week 18 | 66.7 [30.8 to 87.0] | 46.2 [17.9 to 70.7]
  >100 kg Week 20: number analyzed (Participants) | 12 | 13
  >100 kg Week 20 | 66.7 [30.8 to 87.0] | 46.2 [17.9 to 70.7]
  >100 kg Week 22: number analyzed (Participants) | 12 | 13
  >100 kg Week 22 | 75.0 [35.5 to 92.3] | 46.2 [17.9 to 70.7]
  >100 kg Week 24: number analyzed (Participants) | 12 | 13
  >100 kg Week 24 | 75.0 [35.5 to 92.3] | 53.8 [23.1 to 77.0]
  >100 kg Week 26: number analyzed (Participants) | 12 | 13
  >100 kg Week 26 | 75.0 [35.5 to 92.3] | 53.8 [23.1 to 77.0]
  >100 kg Week 28: number analyzed (Participants) | 12 | 13
  >100 kg Week 28 | 75.0 [35.5 to 92.3] | 53.8 [23.1 to 77.0]

4. Secondary Outcome: Having PASI 100 Response, Assessed Separately at Weeks 4, 8, and 28.
Description: Having 100% improvement from baseline in PASI score. The outcome measure is summarized using the least squares mean percentage of subjects having PASI 100 response at Weeks 4, 8, and 28, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline PASI score.
  The PASI is the most widely used tool in clinical practice and clinical trials to assess psoriasis severity and extent. Assessment is done based on the condition of the disease at the time of evaluation, not in relation to the condition at a previous visit. The investigator assesses the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions (head/neck, trunk, upper extremities, lower extremities) according to a severity scale. The investigator also assesses the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe/extensive condition.
Time Frame: Weeks 4, 8, and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of participants
  Week 4 | 23.3 [12.0 to 34.6] | 1.9 [-1.8 to 5.6]
  Week 8 | 40.8 [27.5 to 54.1] | 16.5 [6.5 to 26.4]
  Week 28 | 61.4 [48.3 to 74.5] | 36.8 [23.9 to 49.8]

5. Secondary Outcome: Having PASI 90 Response, Assessed Separately at Weeks 4, 8, 16, and 28.
Description: Having 90% improvement from baseline in PASI score. The outcome measure is summarized using the least squares mean percentage of subjects having PASI 90 response at Weeks 4, 8, 16, and 28, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline PASI score.
  The PASI is the most widely used tool in clinical practice and clinical trials to assess psoriasis severity and extent. Assessment is done based on the condition of the disease at the time of evaluation, not in relation to the condition at a previous visit. The investigator assesses the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions (head/neck, trunk, upper extremities, lower extremities) according to a severity scale. The investigator also assesses extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe/extensive condition.
Time Frame: Weeks 4, 8, 16, and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of participants
  Week 4 | 28.7 [16.7 to 40.8] | 9.2 [1.4 to 16.9]
  Week 8 | 60.2 [46.8 to 73.7] | 24.9 [13.1 to 36.7]
  Week 16 | 69.1 [56.7 to 81.5] | 45.2 [31.8 to 58.6]
  Week 28 | 69.8 [57.4 to 82.2] | 44.7 [31.2 to 58.2]

6. Secondary Outcome: Having Investigator's Global Assessment (IGA) of 0, Assessed Separately at Weeks 16 and 28.
Description: Having a score of 0 (clear) in IGA. The outcome measure is summarized using the least squares mean percentage of subjects having an IGA score of 0 at Weeks 16 and 28, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline IGA score.
  The IGA is an instrument used in clinical trials to rate the severity of psoriasis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Weeks 16 and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of participants
  Week 16 | 55.5 [42.3 to 68.7] | 35.6 [22.8 to 48.3]
  Week 28 | 62.4 [49.5 to 75.3] | 41.2 [28.1 to 54.3]

7. Secondary Outcome: Having IGA of 0 or 1, Assessed Separately at Weeks 16 and 28.
Description: Having a score of 0 (clear) or 1 (almost clear) in IGA. The outcome measure is summarized using the least squares mean percentage of subjects having an IGA score of 0 or 1 at Weeks 16 and 28, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline IGA score.
  The IGA is an instrument used in clinical trials to rate the severity of psoriasis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Weeks 16 and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of participants
  Week 16 | 78.5 [67.5 to 89.5] | 52.5 [39.1 to 66.0]
  Week 28 | 82.1 [71.8 to 92.4] | 65.4 [52.7 to 78.2]

8. Secondary Outcome: Having Dermatology Life Quality Index (DLQI) Total Score of 0 or 1, Assessed Separately at Weeks 4, 8, 12, 16, 20, 24, and 28.
Description: The outcome measure is summarized using the least squares mean percentage of subjects having a DLQI score of 0 or 1 at Weeks 4, 8, 12, 16, 20, 24, and 28, based on a logistic regression model adjusted for baseline body weight (<=100 kg,>100 kg) and baseline DLQI score.
  The DLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all/not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
percentage of participants
  Week 4 | 67.8 [54.9 to 80.8] | 34.3 [21.1 to 47.6]
  Week 8 | 68.8 [56.2 to 81.3] | 66.8 [53.7 to 79.8]
  Week 12 | 78.4 [66.8 to 89.9] | 66.0 [52.7 to 79.2]
  Week 16 | 80.2 [69.7 to 90.8] | 71.6 [59.7 to 83.4]
  Week 20 | 80.0 [69.0 to 90.9] | 68.9 [56.3 to 81.4]
  Week 24 | 75.7 [64.0 to 87.3] | 70.6 [58.3 to 82.9]
  Week 28 | 79.3 [68.3 to 90.3] | 66.6 [53.9 to 79.3]

9. Secondary Outcome: Change in 36-Item Short Form Health Survey Version 2 (SF-36v2) Physical Component Score From Baseline, Assessed Separately at Weeks 4, 8, 16, and 28.
Description: The SF-36v2 is a 36-item general health status assessment. Participants answer each question by selecting 1 of 3 to 6 categorical response options. The SF-36v2 yields scores for 8 health domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) and 2 psychometrically derived summary scores (a physical component summary and a mental component summary). The physical component summary score ranges from 5.1 to 79.7. Higher scores indicate better outcome.
Time Frame: Weeks 4, 8, 16, and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
score on a scale
  Week 4 | 3.3 [1.9 to 4.7] | 1.9 [0.4 to 3.3]
  Week 8 | 3.8 [2.5 to 5.1] | 3.0 [1.6 to 4.4]
  Week 16 | 4.2 [2.7 to 5.6] | 3.7 [2.2 to 5.1]
  Week 28 | 3.9 [2.5 to 5.3] | 3.9 [2.5 to 5.3]

10. Secondary Outcome: Change in 36-Item Short Form Health Survey Version 2 (SF-36v2) Mental Component Score From Baseline, Assessed Separately at Weeks 4, 8, 16, and 28.
Description: The SF-36v2 is a 36-item general health status assessment. Participants answer each question by selecting 1 of 3 to 6 categorical response options. The SF-36v2 yields scores for 8 health domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) and 2 psychometrically derived summary scores (a physical component summary and a mental component summary). The mental component summary score ranges from -4.0 to 79.7. Higher scores indicate better outcome.
Time Frame: Weeks 4, 8, 16, and 28
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
score on a scale
  Week 4 | 2.7 [1.3 to 4.1] | 2.6 [1.2 to 4.0]
  Week 8 | 3.8 [2.3 to 5.2] | 3.7 [2.2 to 5.2]
  Week 16 | 3.0 [1.5 to 4.4] | 3.6 [2.1 to 5.1]
  Week 28 | 3.1 [1.3 to 4.9] | 4.0 [2.2 to 5.8]

11. Secondary Outcome: Occurrence of Treatment-emergent Adverse Events (AEs) From Baseline to Week 28.
Description: An adverse event is considered treatment-emergent if the onset occurred after the first administration of IMP or if the event started prior to the first administration of IMP and worsened in severity after the first administration of IMP.
Time Frame: From baseline to Week 28
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
Number analyzed (Participants) | 56 | 56
Participants | 42 | 31

ADVERSE EVENTS:
Time Frame: 28 Weeks
Description: Treatment-emergent adverse events
Arm/Group | Arm 1 (Brodalumab + Dummy 1) | Arm 2 (Guselkumab + Dummy 2)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 4/56 | 4/56
Other Adverse Events (participants affected / at risk) | 37/56 | 25/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Brodalumab + Dummy 1) (N=56) | Arm 2 (Guselkumab + Dummy 2) (N=56)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Brodalumab + Dummy 1) (N=56) | Arm 2 (Guselkumab + Dummy 2) (N=56)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (14) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 6 (6)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 5 (10) | 3 (4)
Depression (Psychiatric disorders) | 3 (3) | 5 (5)
Hypertension (Vascular disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all phase 3 clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT04533737/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04533737/SAP_001.pdf